CLINICAL TRIAL: NCT06434883
Title: Assessment of an App-based Anxiety/Depression Program in a Population With Elevated Anxiety/Depression A Clinical Randomized Controlled Trial
Brief Title: Assessment of an App-based Anxiety/Depression Program in a Population With Elevated Anxiety/Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Ulrich Kirk, Associate Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 434587
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Depression Anxiety Disorder
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anxiety/Depression Program (Active Comparator)
  Interventions: Behavioral: Anxiety/Depression Program
- Waitlist (Other)
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: Anxiety/Depression Program — Participants will complete the Headspace Anxiety/Depression Program, which is a 21 day program based on CBT, combined with mindfulness. The program is trans-diagnostic in nature (i.e. addresses both anxiety and depression symptoms).
  Arms: Anxiety/Depression Program
Other: Waitlist — Participants will continue their regular routines for an 21 day period and will not be assigned to an intervention.
  Arms: Waitlist

SUMMARY:
Generalized anxiety disorder is a mental health disorder characterized by feelings of tension and worry with physical symptoms including increased blood pressure. Approximately 20% of US adults reported an anxiety disorder in the past year and an estimated 31% of US adults reported anxiety at some time in their lives. Anxiety can be experienced throughout one's life and levels of anxiety can increase with stressful life events, physical health conditions, and medication use. Chronic, untreated anxiety has been linked to headaches, dizziness, depression, high blood pressure, heart disease, digestive disorders, and a worsened immune system - greatly impacting one's overall quality of life (QOL).

Anxiety and depression are highly comorbid, with approximately 50-60% of those with anxiety symptoms also experiencing depression symptoms. Experiencing these disorders and symptoms comorbidly may further worsen one's mental health and overall QOL. Untreated, chronic depression can heighten symptoms of depression leading to increased risk of heart disease, sleep disruptions, weight gain/loss, a weakened immune system, physical pains, and suicide attempts.

Anxiety and depression are commonly treated using various psychotherapeutic techniques including cognitive behavioral therapy (CBT) and acceptance and commitment therapy techniques administered by a licensed therapist. However, therapy has many barriers to treatment including insurance not covering treatments, overall treatment cost, unsure where to seek treatment/no access to a therapist, and therapy being unavailable and inconvenient due to scheduling during the workday. As such, app-based mental health tools have increased in popularity to improve access and affordability to effective mental health treatments.

The purpose of the study is to examine the effectiveness of a guided anxiety/depression app-based program by Headspace, which uses CBT with mindfulness to improve anxiety and depression symptoms in a population with elevated baseline anxiety and/or depression. The study will employ a 2-arm app-based intervention involving 1 active intervention and a waitlist control for a duration of 3 weeks, followed by a 3-week follow-up assessment.

DETAILED DESCRIPTION:
Participants who meet the inclusion criteria will complete the informed consent procedure and the baseline assessment consisting of the study's primary outcomes of anxiety (GAD-7) and depression (PHQ-8) and the secondary outcome measures including sleep quality using the PSQI, perceived stress using the PSS-10, mindfulness using the MAAS, well-being using the WEMWBS, and report use of prescription medication. After the baseline assessment, participants will be randomized into one of two groups (Headspace Anxiety/Depression Program or waitlist control). Participants will participate in the intervention/waitlist control group for 3 weeks. Having completed the 3 week intervention, participants will complete the post-intervention assessment consisting of the primary and secondary outcome measures. Finally, participants will complete the follow-up assessment 3 weeks after post-intervention with a questionnaire to assess changes in routines (including physical activity, prescription medication use or treatments), and the primary and secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of anxiety (defined as a score of 10 or greater on the GAD-7) and/or depression (defined as a score of 10 or greater on the PHQ-8).
* Prescription medication for anxiety, depressive symptoms provided a stable dose for ≥4 weeks before baseline or no medication.
* 18+ years old.
* Based in the U.S.
* Access to a smartphone device, as the intervention will be delivered via a smartphone application.

Exclusion Criteria:

* A diagnosis of any of the following conditions: self-reported schizophrenia, psychosis, bipolar disorder, seizure disorder, substance use disorder, recent trauma to the head or brain damage, severe cognitive impairment, serious physical health concerns necessitating surgery or with a prognosis of less than 6 months, or pregnancy.
* Not being on a stable dose of anxiety or depression medication for ≥4 weeks.
* Risks associated with suicidal ideation and risk of self-harm.
* Two or more hospitalizations within the past 6 months for psychiatric reasons.
* Completed CBT (or another "active" form of psychotherapy that includes self-monitoring and cognitive and/or behavioral exercises) delivered by a licensed therapist in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-8 (PHQ8) | Change from baseline to immediately post-intervention and 3-week follow-up
  The PHQ-8 is used to measure depression symptoms. The PHQ-8 consists of 8 items. Participants use a Likert scale ranging from 0 = not at all to 3 = nearly every day. The range of PHQ-8 scores is 0-24.
General Anxiety Disorder-7 (GAD-7) | Change from baseline to immediately post-intervention and 3-week follow-up
  The GAD-7 is a 7-item self-report scale based on the Diagnostic and Statistical Manual of Mental Disorders-IV criteria for generalized anxiety disorder, with items scored from 0 (not at all) to 3 (nearly every day).

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to immediately post-intervention and 3-week follow-up
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances. 19 individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Higher scores indicate worse sleep quality where poor sleep will be a PSQI total score of > 5.
Perceived Stress Scale (PSS-10) | Change from baseline to immediately post-intervention and 3-week follow-up
  The PSS is a 10-item scale designed to measure the perception of stress within the past month. Participants use a Likert scale with responses ranging from 0 = never to 4 = very often. PSS-10 scores range from 0-40 with higher scores indicating higher perceived stress. Additionally, scores can be categorized as low (0-13), moderate (14-26), and high (27-40) perceived stress.
Mindful Attention Awareness Scale (MAAS) | Change from baseline to immediately post-intervention and 3-week follow-up
  Mindfulness will be measured by the MAAS. The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness. Each of the 15 items aims at measuring one's awareness of what is taking place at the present. The MAAS is answered on a five-point Likert scale. Higher scores reflect higher dispositional mindfulness.
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Change from baseline to immediately post-intervention and 3-week follow-up
  WEMWBS is a 14 item scale of mental well-being covering subjective well-being and psychological functioning, in which all items are worded positively and address aspects of positive mental health. The scale is scored by summing responses to each item answered on a 1 to 5 Likert scale. The minimum scale score is 14 and the maximum is 70.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Kirk, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data collected in this project will be de-identified and made available on a shared secured data repository. Results from this project will be shared and disseminated, including manuscripts will be written and submitted for publication in peer-reviewed journals/conferences. All necessary ethical approvals will be obtained.
Time Frame: Data will be made available upon request after dissemination of results.

REFERENCES:
- [Background] National Institute of Mental Health (2023). Any Anxiety Disorder. Retrieved April 25, 2023, from https://www.nimh.nih.gov/health/statistics/any-anxiety-disorder.
- [Background] American Psychological Association (2022). Anxiety. Retrieved April 25, 2023, from https://www.apa.org/topics/anxiety.
- [Background] Celano CM, Daunis DJ, Lokko HN, Campbell KA, Huffman JC. Anxiety Disorders and Cardiovascular Disease. Curr Psychiatry Rep. 2016 Nov;18(11):101. doi: 10.1007/s11920-016-0739-5. PMID 27671918
- [Background] Lampl C, Thomas H, Tassorelli C, Katsarava Z, Lainez JM, Lanteri-Minet M, Rastenyte D, Ruiz de la Torre E, Stovner LJ, Andree C, Steiner TJ. Headache, depression and anxiety: associations in the Eurolight project. J Headache Pain. 2016;17:59. doi: 10.1186/s10194-016-0649-2. Epub 2016 Jun 1. PMID 27245683
- [Background] Neuhauser HK. The epidemiology of dizziness and vertigo. Handb Clin Neurol. 2016;137:67-82. doi: 10.1016/B978-0-444-63437-5.00005-4. PMID 27638063
- [Background] Leonard BE, Song C. Stress and the immune system in the etiology of anxiety and depression. Pharmacol Biochem Behav. 1996 May;54(1):299-303. doi: 10.1016/0091-3057(95)02158-2. PMID 8728571
- [Background] Saha L. Irritable bowel syndrome: pathogenesis, diagnosis, treatment, and evidence-based medicine. World J Gastroenterol. 2014 Jun 14;20(22):6759-73. doi: 10.3748/wjg.v20.i22.6759. PMID 24944467
- [Background] National Alliance on Mental Illness (2018). The Comorbidity of Anxiety and Depression. Retrieved April 25, 2023, from https://www.nami.org/blogs/nami-blog/january-2018/the-comorbidity-of-anxiety-and-depression.
- [Background] Hirschfeld RM. The Comorbidity of Major Depression and Anxiety Disorders: Recognition and Management in Primary Care. Prim Care Companion J Clin Psychiatry. 2001 Dec;3(6):244-254. doi: 10.4088/pcc.v03n0609. PMID 15014592
- [Background] Andrade LH, Alonso J, Mneimneh Z, Wells JE, Al-Hamzawi A, Borges G, Bromet E, Bruffaerts R, de Girolamo G, de Graaf R, Florescu S, Gureje O, Hinkov HR, Hu C, Huang Y, Hwang I, Jin R, Karam EG, Kovess-Masfety V, Levinson D, Matschinger H, O'Neill S, Posada-Villa J, Sagar R, Sampson NA, Sasu C, Stein DJ, Takeshima T, Viana MC, Xavier M, Kessler RC. Barriers to mental health treatment: results from the WHO World Mental Health surveys. Psychol Med. 2014 Apr;44(6):1303-17. doi: 10.1017/S0033291713001943. Epub 2013 Aug 9. PMID 23931656
- [Background] Centers for Disease Control and Prevention (2018). Prevalence of Depression Among Adults Aged 20 and Over: United States, 2013-2016. Retrieved April 25, 2023, from https://www.cdc.gov/nchs/products/databriefs/db303.htm.
- [Derived] Staiano W, Callahan CE, Davis M, Tanner L, Kunkle S, Glover J, Kole J, Bakshi N, Romagnoli M, Kirk U. Efficacy of a Self-Guided Transdiagnostic Intervention for Adults With Anxiety and Depression: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Oct 23;13:e79759. doi: 10.2196/79759. PMID 41129814